CLINICAL TRIAL: NCT06892847
Title: Brain STimulation for ANxiety and Depression in Youth: Brain STAND
Brief Title: Brain STimulation for ANxiety and Depression in Youth
Acronym: Brain STAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Kara Murias, Assistant Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB25-0288
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Magnetic Stimulation (TMS) (Experimental): Open-label study with active TMS for treatment.
  Interventions: Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — Participants will receive TMS for treatment measures as determined by referral and presentation.
  Other Names: TMS

SUMMARY:
In this open-label trial, the overall aim is to determine if TMS treatment can improve anxiety and depression in a broad group of children and youth referred by physicians.

DETAILED DESCRIPTION:
Mental health disorders are a leading cause of disability, and approximately 14% of adolescents are diagnosed globally. Within Canada, the prevalence of mental health disorders is increasing, with youth aged 15-24 years being greatly impacted. Broadly, mental health disorders include anxiety, post-traumatic stress disorders, depression, schizophrenia, disruptive behaviour, and neurodevelopmental disorders such as autism spectrum disorder (ASD), and attention-deficit/hyperactivity disorder (ADHD). Mental health disorders are associated with clinically significant disrupted behaviour, emotional regulation, and thinking, and can limit one's ability to participate in activities of daily living and drastically impact quality of life. Moreover, a variety of negative outcomes can be associated with these mental health disorders, including health and development-related concerns regarding educational achievement, substance abuse, violence, reproductive and sexual health. In Canada, suicide was the fourth leading cause of death in children (age 1-14; after cancer, accidental injuries and congenital malformations) and the second leading cause of death in youth (age 15-19; after accidental injury) in 2023 according to Stats Can. https://www150.statcan.gc.ca/.

The literature suggests the peak age of mental health disorder onset within the general global population is 14.5 years; a recent meta-analysis of 192 epidemiological studies also reported approximately 83% of individuals with neurodevelopmental disorders experienced onset by the age of 18 years. Further, approximately 52% of individuals with anxiety or fear-related disorders, 48% with feeding or eating disorders or problems, 45% with obsessive-compulsive or related disorders, 28% with stress disorders, and 12% with mood disorders experienced onset by the age of 18 years. The high prevalence of mental health disorders within the child and youth population, and the limited options and availability of therapy choices is contributing to the need to explore additional treatment opportunities.

Interventions for mental health disorders commonly include psycho-social and pharmacological approaches, though these therapies are largely modelled after adult populations, with some indication that medications are not as effective in children and adolescents. Pharmacotherapy may be accompanied by side-effects, and adverse experiences with psychotropic medications at a young age reportedly contribute to poor long-term adherence to other psychiatric therapies. Many families and patients have strong preference for nonpharmaceutical treatments, which can limit options. Another proposed intervention strategy for mental health disorders involves non-invasive brain stimulation, including transcranial magnetic stimulation (TMS). TMS elicits changes in neural population activation with the use of repetitive TMS (rTMS) or theta-burst stimulation. TMS has been used for the treatment of anxiety and depression in adults, and both TMS and TBS have been well-tolerated in children, with only mild transient side effects noted. TMS may be an effective adjunct or sole treatment for mental health disorders in youth; for example, when combined with antidepressants, rTMS increased the treatment effect in 8-24-year-olds with depression, and therefore the clinical application of TMS for mental health disorders in youth requires further investigation. In the United States, rTMS has been approved for the treatment of depression in adolescents starting at the age of 15, and there are encouraging results in implementation studies in other jurisdictions. To ensure adolescents in Canada have access to this therapy, clinical care pathways (such as appropriate referral criteria, outcome measures, and resource requirements) must be better understood.

There are indications that TMS is effective and safe in many populations that are at high risk of depression. For example, TMS has shown to be safe and effective for treatment of depression during pregnancy. In contrast, the use of antidepressants during pregnancy is associated with a risk (though low) of adverse effects for both mother and fetus. Furthermore, treatment of anxiety and depression in complex populations with co-occurring conditions, such as in patients with neurodevelopmental disorders, has limited research in general and in neurostimulations specifically. Despite the recent approval in the United States, evidence for neurostimulation in children and adolescents is lagging behind that of adults. Given the burden of disease in this population, improvement in research, particularly implementation and clinical integration, is both a clinical and ethical imperative.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 6 and 18 years old
2. diagnosis of anxiety or depression made by a qualified medical professional
3. active anxiety and/or depression symptoms

Exclusion Criteria:

1. status epilepticus in past 12-months
2. presence of any disease, medical condition, or physical condition that, in the opinion of the study investigator may compromise, interfere, limit, affect, or reduce the participant's ability to complete the study
3. hospitalization for suicide attempt within the past 3 months (unless participant is under the daily supervision of a physician, such as in a mental health day treatment program)
4. TMS-related contraindications, including implanted medical devices (e.g., pacemaker)
5. if actively taking prescription medication, no changes in medication for at least 3 months prior to entry into the study, with no anticipation of change in the frequency or dose over the duration of the study, unless changes to medication are required for participant safety
6. unable to understand instructions in English

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Revised Children Anxiety and Depression Scale (RCADS) | Baseline and 5 weeks.
  This 47-item questionnaire assesses the presence and severity of anxiety and depression symptoms. Items are rated from 0 (never) to 3 (always) and includes six subscales, with higher total scores indicating greater severity of symptoms.

SECONDARY OUTCOMES:
Children's Global Assessment Scale (CGAS) | Baseline and 5 weeks.
  This physician-rated scale assesses medical history, symptoms, behaviour, and psychosocial circumstances to determine level of general functioning. A score is entered from 100 (superior functioning) to 0 (needs constant supervision).
PROMIS Pain Interference-8a | Baseline and 5 weeks.
  This 8-item questionnaire assesses the impact of pain on aspects of daily living in the past 7 days. Items are rated from 0 (never) to 4 (almost always), with higher scores indicating pain has a greater impact on activities of daily life.
Pediatric Quality of Life Inventory (PedsQL) | Baseline and 5 weeks
  This 28-item questionnaire assesses health-related quality of life in the past month. This tool evaluates multiple domains, including physical, emotional, social, and school functioning. Items are rated from 0 (never) to 4 (almost always), with lower scores indicating greater quality of life.
Emotional Dysregulation Inventory (EDI) short form | Baseline and 5 weeks.
  This 13-item questionnaire evaluates emotional dysregulation in the past 7 days. This tool is scored from 0 (not at all) to 4 (very severe), with greater scores indicating more emotional dysregulation.
Youth Life Interference Scale (YLIS) | Baseline and 5 weeks.
  This 11-item questionnaire assesses the impact of mental health symptoms on daily life in the past 2 weeks. Items are rated from 0 (not at all) to 4 (a great deal), with lower scores indicating mental health symptoms had less impact on daily life.
Pubertal Development Scale (PDS) | Baseline
  This 5-item questionnaire is used to determine an individual's puberty development category, including pre-pubertal, early pubertal, mid-pubertal, late pubertal, post-pubertal.
Early Psychosis Screener-26 (EPS-26) | Baseline
  This 26-item questionnaire assesses symptoms of psychosis, including hallucinations and delusions, in the past 30 days. Items are rated from 1 (never) to 5 (always), with lower scores indicating fewer symptoms of psychosis.
Strengths and Weaknesses of Attention-Deficit/Hyperactivity Disorder and Normal Behaviour Scale (SWAN) | Baseline and 5 weeks.
  This 30-item questionnaire assesses strengths and difficulties with attention and behaviour regulation. This questionnaire compares attention, activity, and impulse to others of similar age, using a scale ranging from far below to far above average.
Aberrant Behavioural Checklist (ABC) | Baseline and 5 weeks.
  This 58-item questionnaire assesses behaviour in the past 4 weeks, using a scale from 0 (not at all a problem) to 3 (the problem is severe in degree). This questionnaire includes 5 domains: irritability, hyperactivity, social withdrawal, stereotypic behaviour, and inappropriate speech.
NIH Toolbox Cognition Battery | Baseline and 5 weeks.
  This battery assesses attention, executive function, and memory and will be completed in-person on a tablet. Specifically, the List Sorting Working Memory Test, Dimension Change Card Sort Test, Flanker Inhibitory Control and Attention Test, and Picture Sequence Memory Test will be administered and take less than 20 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Murias, MD/PhD, Principal Investigator — The University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No